CLINICAL TRIAL: NCT05531370
Title: Implementation of Evidence-based Breathing Retraining for Patients with Asthma in Region Zealand, Denmark
Brief Title: Implementation of Evidence-based Breathing Retraining for Patients with Asthma in Region Zealand
Acronym: EmBRAiZ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMN-2022-01229
Record Dates: First submitted 2022-07-04; First posted 2022-09-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: Implementation; Asthma; Breathing Retraining
MeSH Terms: conditions — Asthma | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breathing Retraining (BR) (Experimental): Patients will receive three sessions (60 min, 30 min, 30 min) of breathing retraining (BR), 1-to-1 with a trained physiotherapist.
  As preferred by the patient:
  * Hybrid delivery mode of BR (H-BR): First session on-site at hospital/clinic for initial assessment and introduction, and following sessions online (MedComs VDX platform or equal; participants access using web cam and sound on smart phone, tablet, or pc).
  * Ordinary delivery of BR: Three sessions on-site at hospital/clinic.
  Interventions: Other: Breathing Retraining

INTERVENTIONS:
Other: Breathing Retraining — Conforming the real-world setting, all participants will continue standard asthma care, i.e., acute and planned visits at GP or pulmonologist.
  BR aims to normalize the inhaled volume, nasal inhalation, exhalation to the resting position of the chest (functional residual capacity, FRC), use of the diaphragm muscle, and to move lower parts of the chest in a frequency of 12-16 per minute. This pattern is initially trained in rest (e.g., side lying or sitting), then during physical activity (e.g., walking). Uncontrolled coughing, frequent yawning or sighing is handled by a suppression technique. Relaxation technique is introduced as a separate activity but to be combined with the breathing pattern method to be used in both resting and as possible during physical activity.
  Other Names: Breathing Exercises

SUMMARY:
This study aims to implement the evidence-based intervention breathing retraining into clinical care of patients with symptomatic asthma irrespective of asthma severity or comorbidities, and in a diverse multicentre setting to evaluate implementation outcomes. This will meet patients' needs and improve health and life situation in patients with uncontrolled asthma. Further, the study will evaluate implementation outcomes.

DETAILED DESCRIPTION:
This study is a hybrid-designed prospective multicenter implementation evaluation study, in which the investigators secondarily will maintain measuring effectiveness of breathing retraining in a real-world setting including primary and secondary health care and add cross-sectorial co-operation. Thus, investigators include more primary outcomes.

The study is part of Exercise First-project, a collaboration of The National Health Service, Region Zealand and the research unit PROgrez, Department of Physiotherapy and Occupational Therapy at Næstved, Slagelse, Ringsted hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma;
* Incompletely controlled asthma or worse: Asthma Control Questionnaire (ACQ5) score ≥0.8;
* Residence (or asthma treatment program) in Region Zealand, Denmark;
* Able to read and understand Danish or available assistance to help understand information material, intervention content and respond to questionnaires.

Exclusion Criteria:

* Unwilling to participate;
* Unable to participate in the intervention due to physical or mental condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of intervention (Uptake) | Through study completion, an average of 1 year
  Organization-related (Pulmonologists, general practioners, physiotherapists) outcome: Proportion of general practices and of hospitals that will adopt BR.
Implementation of intervention (Fidelity) | Through study completion, an average of 1 year
  Organization-related (physiotherapists) outcome:
  % of contents delivered as planned assessed by a checklist of key aspects in the breathing retraining-intervention.
Feasibility of online sessions in Hybrid delivery mode of BR (H-BR) (Acceptability) | Through study completion, an average of 1 year
  Patient- and Organization-related (physiotherapists) outcome: assessed by a semi-structured interview.
Effectiveness: MiniAsthma Quality of Life Questionnaire, MiniAQLQ | Through study completion, an average of 1 year
  Patient-related outcome, disease specific quality of life questionnaire. 7-point Likert scales from 1-7, 1 = worse outcome, 7 = better outcome.
  Success rates of improvements minus deteriorations of individual effects, measured at 12 month follow up.

SECONDARY OUTCOMES:
MiniAsthma Quality of Life Questionnaire, MiniAQLQ | Change from baseline to 12 months
  Patient-related outcome: Mean of disease specific quality of life questionnaire. 7-point Likert scales from 1-7, 1 = worse outcome, 7 = better outcome.
Breathing pattern observation | Change from baseline to 12 month
  Patient-related outcome. Pre-defined key aspects of the breathing pattern assessed qualitatively observation by the physiotherapist.
Objective physical activity level | Change from baseline to 12 month
  Patient-related outcome. Objectively measured physical activity and inactivity using combined wearable thigh and wrist accelerometers, worn for seven consecutive days.
Objective steps per day (average) | Change from baseline to 12 month
  Patient-related outcome. Objectively measured steps per day using combined wearable thigh and wrist accelerometers, worn for seven consecutive days.

OTHER OUTCOMES:
Ashma severity by Global Initiative for Asthma (GINA) treatment steps | Change from baseline to 12 month
  Patient-related outcome. Asthma severity assessed by pharmacotherapy level, calculated into GINA treatment steps 1-5 (1 = mild asthma, 5 = severe asthma), using a questionnaire completed by the physiotherapist during an interview with the patient.
Adverse events (Safety) | Post-intervention (3-month)
  Patient-related outcome; number, % caused discontinuation.
Asthma Control Questionnaire, ACQ5 | Change from baseline to 12 month
  Patient-related outcome: ACQ5 i.e. item 1-5 of the ACQ. Mean of asthma symptom level questionnaire; 7-point Likert scales from 0-6, 0 = better outcome, 6 = worse outcome.
Number of online sessions delivered | Post-intervention (3-month)
  Number, % of total sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Søren T Skou, Prof., Study Chair — Naestved-Slagelse-Ringsted Hospitals; University of Southern Denmark; Lars H Tang, Assoc.Prof., Study Chair — Naestved-Slagelse-Ringsted Hospitals; University of Southern Denmark; Cecilie L Egholm, PostDoc., Study Chair — Naestved-Slagelse-Ringsted Hospitals, Denmark; Uffe Bodtger, Prof., Study Chair — Zealand University Hospital; University of Southern Denmark; Mike Thomas, Prof., Study Chair — Primary Care Research University of Southampton, UK; Karen H Andreasson, Dr., Principal Investigator — Naestved-Slagelse-Ringsted Hospitals; University of Southern Denmark
Locations (1):
- Naestved Hospital, Næstved, Region Sjælland, Denmark